CLINICAL TRIAL: NCT02672540
Title: A Phase II, Multicenter, Single-Blind, Randomized Study of the Safety and Effectiveness of SANGUINATE™ Versus Normal Saline in Adult Sickle Cell Disease Patients With Vaso-Occlusive Crisis (VOC)
Brief Title: A Study of SANGUINATE for the Treatment of Vaso-occlusive Crisis (VOC) in Adult Sickle Cell Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGSC-002
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell; Anemia; VOC; Vaso occlusive crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Vaso-Occlusive Crises | interventions — PEGylated carboxyhemoglobin bovine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SANGUINATE 320 mg/kg (Experimental): Two-hour infusion of SANGUINATE on Day 1 and Day 2
  Interventions: Drug: SANGUINATE 320 mg/kg
- Normal Saline (Placebo Comparator): Two-hour infusion of Normal Saline and Day 1 and Day 2
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: SANGUINATE 320 mg/kg — Two-hour infusion of SANGUINATE on Day 1 and Day 2
  Other Names: pegylated carboxyhemoglobin bovine
  Arms: SANGUINATE 320 mg/kg
Drug: Normal Saline — Two-hour infusion of Normal Saline and Day 1 and Day 2
  Arms: Normal Saline

SUMMARY:
Safety and effect of SANGUINATE on Sickle Cell Disease patients experiencing a vaso-occlusive crisis who are admitted to the hospital for treatment.

DETAILED DESCRIPTION:
A single-blind, multicenter, randomized, placebo-control study in which 30 Sickle Cell disease patients having a vaso-occlusive crisis will either receive SANGUINATE 320 mg/kg/patient (8 mL/kg/patient) or Normal Saline on Day 1 (Visit 1) and Day 2 (Visit 2) infused over 2 hours each day. Patients are to remain in the hospital for up to 7 days but can be discharged at any time after receiving the second dose of SANGUINATE, provided their vaso-occlusive crisis has resolved and the patient has completed discharge procedures. Patients will have a follow-up phone call 7 days after discharge from the hospital to obtain safety, concomitant medication and pain assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 65 years of age
2. Diagnosis of Sickle Cell Disease (Hb-SS or any Genotype)
3. Pain-score due to vaso-occlusive pain crisis (VOC) ≥ 8 on a 10 point scale
4. VOC pain location ≥ 1 sites typical of vaso-occlusive crisis
5. Patients with Priapism, acute chest syndrome, and/or with other Sickle Cell Disease comorbidities can be enrolled with good judgment of the Investigator.
6. Signed and dated informed written consent by the subject
7. Able to receive intravenous infusion of SANGUINATE or Normal Saline
8. Women of childbearing potential with a negative serum pregnancy test and using a reliable method of contraception during the study period and for 30 days thereafter. Male study participants also agree to use contraception for 30 days after the study period

Exclusion Criteria:

1. In the judgment of the investigator, the patient is not a good candidate for the study
2. Females who are lactating and/or breastfeeding
3. Fewer than 14 days since prior infusion pain medication treatment for VOC
4. Medical history or evidence of moderate to severe renal insufficiency (estimated GFR < 60 mL/min) or chronic kidney disease, or of moderate to severe hepatic disease (ALTs > 5 x ULN)
5. Concurrent or prior treatment within 30 days of Screening with an investigational medication.
6. Symptoms or electrocardiogram (ECG)-based signs of acute myocardial infarction, unstable angina pectoris, decompensated heart failure, third degree heart block or cardiac arrhythmia associated with hemodynamic instability;
7. Severe or unstable concomitant condition or disease (e.g., known significant neurologic deficit, cancer, hematologic, metabolic or coronary disease), or chronic condition (e.g., psychiatric disorder), that, in the opinion of the Investigator, may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results;
8. Evidence or history of regular alcohol abuse
9. Screening laboratory result indicating serologic positivity for hepatitis C antibodies or hepatitis B surface antigens, unless explained by a documented vaccination.
10. Unable to comply with study attendance, protocol procedures or other study requirements;
11. Abnormal Echocardiogram at Study Entry (defined as Tricuspid Regurgitant Jet Velocity >3.1 m/sec).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Time to readiness for discharge from in hospital stay following treatment with SANGUINATE and Normal Saline. | Up to 7 Days
  Defined as the patient's response that their pain episode has improved enough for discharge from the hospital, or the Investigator's assessment that the patient is ready for discharge from the hospital.

SECONDARY OUTCOMES:
Safety of treatment as defined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis measures, as well as reported increases in pain and other reported adverse events | Up to 7 Days
  Composite endpoint with multiple vital signs, ECGs, echocardiograms, clinical assessments and bio-analytical lab measurements over the 7 day time frame
Proportion of patients who develop acute chest syndrome (ACS) during the study. | Up to 14 Days
Proportion of patients who are re-hospitalized for their vaso-occlusive crisis episode. | Up to 7 Days
Total length of stay (LOS) following treatment of SANGUINATE versus Normal Saline. | Up to 7 Days
Percent reduction in total pain medication required during in-hospital stay following treatment with SANGUINATE and Normal Saline. | Up to 7 Days
Percent reduction in pain score utilizing a visual analog scale following treatment with SANGUINATE and Normal Saline. | Up to 7 Days
Reduction in the level of C-Reactive Protein following treatment of SANGUINATE versus Normal Saline. | Up to 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Misra, PhD, Study Director — Prolong Pharmaceuticals
Locations (4):
- Bogotá, Colombia
- Santo Domingo, Dominican Republic
- San Pedro Sula, Honduras
- Panama City, Panama

IPD SHARING:
Plan to Share IPD: No